CLINICAL TRIAL: NCT06500429
Title: A Proof-of-Concept, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety and Efficacy of Oral NG101 in the Treatment of Side Effects in Healthy Adult Participants Administered a Single Subcutaneous Dose of a Glucagon-Like Peptide 1 Agonist
Brief Title: A Study to Evaluate the Safety and Efficacy of NG101 in Adult Participants Receiving a Glucagon-like Peptide-1 (GLP-1) Agonist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurogastrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NG101-202
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Overweight and Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NG101 20 mg BID (Experimental): NG101 (metopimazine mesylate) 20 mg capsule BID + single SC dose of 0.5 or 1 mg semaglutide
  Interventions: Drug: NG101; Drug: Semaglutide Injectable Product
- Placebo (Placebo Comparator): Placebo capsule BID + single SC dose of 0.5 or 1 mg semaglutide
  Interventions: Drug: Placebo; Drug: Semaglutide Injectable Product

INTERVENTIONS:
Drug: NG101 — NG101 20 mg BID
  Other Names: metopimazine mesylate
  Arms: NG101 20 mg BID
Drug: Placebo — Placebo BID
  Arms: Placebo
Drug: Semaglutide Injectable Product — Semaglutide 0.5 or 1 mg

SUMMARY:
Adult participants with BMI between 22 - 35 kg/m2 will be enrolled and randomized to receive either NG101 (20 mg twice daily [BID]) or placebo for 5 days beginning on Day 1. On Day 2, all participants will receive a single subcutaneous injection of a Glucagon-like Peptide-1 (GLP-1) agonist (semaglutide). Participants will remain at the clinical research unit for the duration of the treatment period.

The goal of this clinical trial is to evaluate the safety and efficacy of NG101 compared to placebo, when also administered along with a GLP-1 agonist, in the management of gastrointestinal side effects commonly associated with GLP-1 agonists for overweight or obesity. Adverse event information will be collected. Gastrointestinal (GI)-specific questionnaires will be used to capture additional details if GI-related adverse events are reported.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Male or female
* BMI between 22 - 35 kg/m2 at screening

Exclusion Criteria:

* Presence or history of illness that might confound the results of the study or pose an -
* History of presence of gastroparesis, gallbladder disease, acute or chronic pancreatitis, or surgery of the abdomen
* History or presence of Type 1 or Type 2 diabetes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Duration of GI-related adverse events | 96 hours following GLP-1 agonist injection
  Number of days with TEAEs of GI-related adverse events following GLP-1 agonist injection
Severity of GI-related adverse events | 96 hours following GLP-1 agonist injection
  Moderate and/or severe TEAES of GI-related adverse events following GLP-1 agonist injection

SECONDARY OUTCOMES:
Number of TEAEs of GI-related adverse events | 96 hours following GLP-1 agonist injection
  Number of TEAEs of GI-related adverse events following GLP-1 agonist injection

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No